CLINICAL TRIAL: NCT04566081
Title: Digital Interventions in Neuro-Rehabilitation (DINR): A Digital Neuro Intervention (DNI) for Word Retrieval (Anomia)
Brief Title: Digital Interventions in Neurorehabilitation: iTALKbetter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18\0071
Record Dates: First submitted 2020-05-29; First posted 2020-09-28 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Aphasia; Anomia
Keywords: Anomia; Word Retrieval; Digital Therapy
MeSH Terms: conditions — Stroke; Aphasia; Anomia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTALKbetter: deterministic (Active Comparator): Participants will receive the deterministic version of the iTALKbetter therapy for 6 weeks. Participants are required to use the therapy for 1.5 hours everyday to reach the required dose of 60 hours over the 6 week period.
  iTALKbetter:deterministic version will randomise the order all of the words that are to be trained and participants will cycle through all of these words regardless of their performance until complete at which point the order is re-randomised and participants begin the cycle again.
  Interventions: Other: iTALKbetter: deterministic
- iTALKbetter: reactive (Active Comparator): Participants will receive the reactive version of the iTALKbetter therapy for 6 weeks. Participants are required to use the therapy for 1.5 hours everyday to reach the required dose of 60 hours over the 6 week period.
  iTALKbetter reactive version is identical to the deterministic version for the first cycle only. From then on the words participants are trained on can change depending on their performance on that word over a number of cycles. Words that participants are failing to retrieve over a number of cycles will be retired from the therapy as they are deemed too difficult for a given participant. Similarly words that are correctly retrieved over a number of consecutive cycles are also retired from the therapy as they are deemed to have been learned. In this way iTALKbetter reactive version will gradually give each participant a personalised corpus of words that they can train on, focusing on the words where they stand to make the most improvements.
  Interventions: Other: iTALKbetter: reactive

INTERVENTIONS:
Other: iTALKbetter: deterministic — A word retrieval therapy application
  Other Names: deterministic iTB
  Arms: iTALKbetter: deterministic
Other: iTALKbetter: reactive — A word retrieval therapy application
  Arms: iTALKbetter: reactive

SUMMARY:
iTALKBetter will provide an app-based therapy for people with word retrieval difficulties who have had a stroke.

This study aims to test the therapy application for people with naming difficulties through a small scale randomized controlled trial.

DETAILED DESCRIPTION:
Mortality from stroke in the UK has reduced from 21% in 1999 to 12% in 2008. However, stroke prevalence has been increasing, the consequence of socioeconomic and scientific advances that have improved survival; which means that more people are surviving with long-standing disability. Language impairment (aphasia) is the second most common major impairment after stroke, with a prevalence of 250,000 in the UK. Aphasia may respond to therapy many months and years after the stroke occurs, but provision of specialist therapy (speech and language therapy - SALT) is far below that needed to provide optimal rehabilitation.

The investigators will address this by targeting a common symptom of post-stroke aphasia: impaired word retrieval problems. This is particularly important in patients receiving rehabilitation for associated disabilities as poor speech production can impair participation/compliance with treatment programmes. The study is designed to improve word retrieval in patients with post-stroke aphasia, who are in the chronic phase (>6 months post-stroke).

The main aim is to test the clinical efficacy of a novel, web-based, DNI. iTALKbetter will provide an effective training tool that patients can use to practice independently. This will free-up SALT time to provide additional assessment, supervision and functional intervention in a highly cost effective manner.

iTALKbetter will provide an app-based therapy for people with word retrieval difficulties who have had a stroke (naming app for a wide variety of common words and phrases).

This Digital Neuro Intervention (DNI) will provide the opportunity for the necessary increased rehabilitation to help people recover lost naming function. This will alleviate NHS Speech and Language Therapist (SALT) time and put users in control of when and where they carry out practice-based language therapy.

Purpose iTALKbetter will provide an app-based therapy for people with word retrieval difficulties who have had a stroke (naming app for a wide variety of common words and phrases).

What does it do? The DNI works via mass practice and feedback to the users on a trial-by-trial basis. The DNI is very simple in a way; it just presents a long series of pictures for users to name. The DNI will use speech recognition (SR) software in order to make a binary decision as to whether the user said the correct word or not. This affects what the next trial (object to name) is and what auditory cue (if any) is provided the next time the user has to name the same item.

What is the clinical trial design? A small, well-defined sample of patients with the potential to benefit from the DNI will be recruited. The main outcome measure is whether the DNI is effective at improving naming impairments. This comparison is within-subject and is achieved by comparing post-therapy measures to multiple baseline measures. A comparison of two different versions of the therapy (a between group comparison) is also planned to answer the secondary question of whether the therapy can be optimised. Outcome measures will be collected by the research team using a variety of standardized and non-standardized tests of language and cognition. These outcome measures are not built into the DNI at this point.

The DNI will be introduced to the participant when attending a testing session. One of the research team will explain how to use the DNI, provide instructions for the user, and give some time for practice items. When confident that the participant can use the DNI independently, the participant will take the device home and continue their therapy (suggested therapy time is 5-10 hours per week) which will be simultaneously monitored by the research team. The research team will also check in on the participant weekly to trouble shoot any difficulties they may have (whether motivational or technical). When the participant has completed the therapy block, they will be invited in again for testing and they will return the mobile device with the DNI on it. The participants who continue to receive standard care during the therapy block will be asked to record and submit details to the research team

Why is the research considered worth doing? Standard (face to face) Speech and Language Therapy (SALT) has a huge evidence-base but patients in the NHS have unmet therapy needs due to a lack of resources. The evidence from speech-therapy highlights the amount of time-on-task required to improve patients' ability to communicate. Naming problems are common and impact on the patients' wellbeing and social inclusion. There is also good evidence that current existing therapeutic approaches work.

A Cochrane review of 39 RCT's involving 2518 participants concluded that speech-therapy results in significant benefits to patients' functional communication. Many of these studies involve high doses of therapy. A meta-analysis examining dose found that positive therapy studies averaged 98 hours of speech therapy in total, while negative studies averaged 43. In the NHS a patient with aphasia can expect a total average of 6-10 hours of SALT. When the intervention takes place or how intensely seems less relevant to recovery. The solution to the lack of available SALT therapy is to produce digital neuro-interventions that give patients the opportunity to practice scientifically validated, impairment based therapy when and where it suits them which gives them access to optimum therapy dose.

Recent improvements in acute stroke care means that demand for already limited NHS resources will increase. Commissioners will need to address this growing unmet need and innovative relatively cheap interventions like this one will provide necessary rehabilitation.

Therapy can be effortful for patients who can sometimes be too fatigued when the therapist comes to do their session. This digital neuro-intervention will provide optimum availability of therapy and therefore place the patient in control of how much they do. The investigators aim to combat this by creating an engaging and adaptive therapy. The adaptiveness will serve to reward the patients for their efforts without ever making them feel like they are failing. This will hopefully boost how long they spend in therapy and therefore make greater gains.

There are therapy 'apps" available for patients with aphasia but the scientific basis for them is lacking and none are targeted for speech production. By using voice recognition software the intervention will be uniquely designed to be used by patients with word retrieval impairments.

What new information will the research provide? The concept of the therapy component is based on standard SALT practice and thus has a strong proof of concept basis, as do the proposed outcome measures. The novel component is packaging it in a user- friendly web-app that is designed for and by people with word-retrieval problems. This is ambitious and yet realistic goal to provide a world-wide evidence-based therapy that can benefit many. This digital neuro-intervention will be in contrast to the plethora of apps available online claiming cognitive training without having scientific proof.

The iTALKbetter research study is a small-scale, randomised, clinical trial for participants with word retrieval impairments post-stroke. The main research question is whether iTALKbetter improves patients' naming ability for trained items. This hypothesis is tested by assessing participants naming abilities on two matched lists of items, half are trained items and half are untrained. A secondary question is whether it matters how the software progresses patients through the therapy. This hypothesis is tested by creating two different versions of iTALKbetter: 'deterministic' and 'reactive'. Participants will be randomised (using minimisation) to one of two of these versions of the therapy. Participants practice with the therapy for set periods of time (therapy block) following a series of (three) baseline measures split over a single, pre-therapy block (see Trial design section 5). The main outcome measure will be a clinically relevant improvement on the naming ability of the trained items (compared to untrained control items). Secondary outcomes include investigating which therapy version optimises recovery on naming accuracy and also improvements in social activity and participation and participant and/or carer reported outcome measures (PROMS).

The investigators also plan to capture brain-based data (structural MRI) in order to test a series of secondary hypotheses relating to both how and why the therapy may work in some participants but not others. All brain imaging will be outside of standard care for the participants and take place at UCL by trained staff.

Hypotheses and Objectives H1-Primary: Does iTB improve naming performance on trained items?

This is a within-subject comparison. The criteria for success is a 10% (raw, or unstandardized) relative improvement in performance. This effect size was used in the recent Big Cactus study.

H2-Secondary: Does reactive iTB significantly improve performance compared with deterministic iTB?

This is two factor analysis with both a within-subject factor (trained vs. untrained items) and a between-group factor (reactive iTB vs. deterministic iTB). The criteria for success is a 5% (raw, or unstandardized) relative difference in performance. This is half the effect size used in the recent Big Cactus study, but that was to compare therapy with no therapy, here expected gains may be more marginal as both groups are receiving the therapy items, just in different orders.

Primary Objective: Does iTB improve naming performance on trained items?

Secondary Objective(s):

The investigators believe that using this DNI will improve word retrieval on trained items by providing a known therapy used by SLT's through a digital app and by enabling an increased dose of therapy. However, another objective is that by using this DNI and practicing every day, there will be changes in participants' brain structure and in the health of the participants and their carers.

* Does reactive iTB significantly improve performance compared with deterministic iTB?
* Are the therapy effects item-specific or do is there generalization to untrained items?
* Are the effects of the DNI therapy limited to the language domain alone or do they improve in other cognitive domains (e.g. sustained attention)?
* Does the DNI improve participant's social activity and participation?
* Is the DNI acceptable to participants (can they use it easily)?
* Is the DNI acceptable to participants' carers?
* Does the DNI improve carer health/well-being?
* Does the DNI have any economic benefits?
* Can baseline structural brain imaging explain participants' responses to the DNI?
* Can baseline structural brain imaging be used to predict incoming participants' response to the DNI?
* Can repeated-measures structural brain imaging identify participants' brain areas that change in response to the DNI?

ELIGIBILITY:
Inclusion Criteria:

* Any type of stroke but at least 6 months after onset.
* Evidence of aphasia on the Comprehensive Aphasia Test
* English as their dominant language
* Able to tolerate MRI brain scan
* Able to give informed consent
* Able to use the DNI (app)

Exclusion Criteria:

* No diagnosis of developmental language disorders
* No diagnosis of severe dementia or primary progressive aphasia
* No major co-existing neurological or psychiatric diagnosis
* No contraindications to brain scanner (e.g. the presence of ferromagnetic implants or other metallic or electronic objects in the body, weight over 24 stone, claustrophobia or pregnancy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Change in accuracy performance on a bespoke Word Retrieval Test: WRT | baseline (week 1), pre intervention (week 12), post-intervention (week 18)
  The WRT is custom test of word retrieval comprised of a subset of the trained and untrained items form the iTALKbetter therapy. Participants accuracy on the word retrieval test is measured at multiple timepoints (baseline, pre intervention, during intervention and post intervention).

SECONDARY OUTCOMES:
Patient and carer reported outcome measures | pre intervention (week 12), post intervention (week 18)
  Qualitative semi-structured interviews to assess a variety of outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P Leff, Professor, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Upton E, Doogan C, Fleming V, Leyton PQ, Barbera D, Zeidman P, Hope T, Latham W, Coley-Fisher H, Price C, Crinion J, Leff A. Efficacy of a gamified digital therapy for speech production in people with chronic aphasia (iTalkBetter): behavioural and imaging outcomes of a phase II item-randomised clinical trial. EClinicalMedicine. 2024 Feb 21;70:102483. doi: 10.1016/j.eclinm.2024.102483. eCollection 2024 Apr. PMID 38685927